CLINICAL TRIAL: NCT00900978
Title: Impact of the 7 Valent Pneumococcal Conjugate Vaccine on Nasopharyngeal Carriage of S. Pneumoniae in Healthy Jordanian Infants.
Brief Title: Impact of the 7 Valent Pneumococcal Conjugate Vaccine (7vPCV) on Nasopharyngeal Carriage of Streptococcus Pneumoniae in Healthy Jordanian Infants
Acronym: 7vPCV
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: German-Jordanian University (Other)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Dr Adnan Al-Lahham, German Jordanian University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0887X1-4611; GPR01703
Record Dates: First submitted 2009-03-16; First posted 2009-05-13 (Estimated); Last update posted 2009-09-30 (Estimated); Status verified 2009-09

CONDITIONS: Streptococcus Pneumoniae
Keywords: Streptococcus pneumoniae; carriage; Resistance; Serotype; vaccination; Colonization of S. pneumoniae
MeSH Terms: interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 7v-PCV (Prevenar) (Experimental): Biological/vaccine
  Interventions: Biological: 7 valent pneumococcal conjugate vaccine (7v-PCV) - Prevenar

INTERVENTIONS:
Biological: 7 valent pneumococcal conjugate vaccine (7v-PCV) - Prevenar — The 7v-PCV will be given to children below 2 years of age. Nasopharyngeal swabs will be taken from the children before vaccination and after finishing the vaccination. The vaccine will be given in a 2+1 scheme.
  Other Names: PREVENAR

SUMMARY:
Nasopharyngeal (NP) colonization of S. pneumoniae in infants is generally acquired at approximately 4-6 months of age. Although there are differences in the prevalence and rank order of serotypes obtained from NP specimens and from those with invasive diseases, pneumococcal nasopharyngeal isolates may reflect the strains circulating in the community and may be used as a marker to predict serotype prevalence of invasive disease and resistance patterns. The information about pneumococcal strains found in Jordanian children and NP-carriage of infants is limited and do not include children living in rural regions. Monitoring serotype distribution is essential for the appropriate application of vaccination. Vaccine use in infants proves to be highly efficacious in the prevention of invasive pneumococcal disease as well as in decreasing the carriage of vaccine serotypes in the nasopharynx of infants which impacted significantly in the long run on otitis media infection and helped decrease the infection rates among contacts of these infants. The result has been a decrease in the pneumococcal infection rate among elderly contacts of these infants and decrease colonization with pneumococci. In order to determine the pneumococcal serotypes which are prevalent among infants attending day care centers (DCCs) in Jordan, a study of these types circulating among infants will be determined over a period of 15 months in 250-300 children attending the DCCs in Ajlun-City by taking 3 NP-swabs, the first before the first vaccine injection in May 2009, the second before the third injection at 10 months of age and the third swab sample is taken at 1 year of age (2-3 months after the last injection with the 7vPCV. The aims of this study were to determine the frequency of NP-carriage and serotype distribution of the strains isolated from infants less than 2 years old, and to get an insight about the coverage of the available and future pneumococcal conjugate vaccines developed for this infectious agent. Good results of this study project would make recommendations for the Ministry of Health (MOH) to include the vaccine in the National Vaccination Program. 15000 doses of the 7v PCV (Prevenar) were donated from Wyeth Pharmaceutical company to the MOH of Jordan in September 2008. These will be vaccinated in a vaccine program (for free) over 15 months period in 2009-2010 in one city in north Jordan called Ajlun. This city has 3676 births per year (Statistics of the MOH 2007). The vaccination program will start from the 18th of May, 2009, and ending in August 2010. The way the vaccine will be given is 2 + 1 injections as recommended by the vaccination committee of the MOH.

DETAILED DESCRIPTION:
S. pneumoniae is one of the major bacterial causes of invasive disease, community acquired pneumonia and respiratory tract infections worldwide (Song, Oh et al. 2008). It causes meningitis, bacteraemia, otitis media, pneumonia and other infections. The resistance rate of this bacteria to antibiotics all over the world is increasing and the mortality rate globally have reached 2 million every year as reported by the WHO. Risk groups are mainly young children under 5 years of age, immune-deficient patients and elderly. There are 91 different serotypes of this infectious agent known worldwide. In the United States of America and Europe, research on S. pneumonia showed that over than 70-85% of all S. pneumoniae cases can be covered and prevented by the 7-valent pneumococcal conjugate vaccine (Prevenar (7v-PCV)). This percentage is different according to the country. In Jordan, this vaccine was introduced and licensed in January 2006 without any previous preliminary studies of the serotypes or capsular types found. Furthermore, there are no published data about the infections caused by Streptococcus pneumonia from Jordan. The total number of Jordanian population is estimated in 2007 to be 5,744 million inhabitants with birth rate 28 per 1000 and these people are concentrated in the capital of Amman (1.781 million), Irbid (629679) and Zarqa (819000). Of Jordanian inhabitants and according to WHO recent numbers of 2008, 37.1% are children below 15 years of age and 3.8% are over than 65 years of age, and total children below 5 years are estimated 2007 to be 917000. This means that the people at risk of pneumococcal infections is 40.9% of the total population. Furthermore, statistical data of the MOH reported an increase of non-meningococcal meningitis cases (without specification of the exact cause of meningitis) from 438 cases (incidence 10.2/ 100,000 population) in 1995 to 778 cases (incidence 14.5/ 100,000 population) in 2007. In 2005, 458 cases/ 747 cases (61%) were from Irbid city alone -north-; and this was 460 cases in 2007 from 778 cases with non meningococcal meningitis. The maximum number of cases with non-meningococcal meningitis was reported in years 2000 (1108 cases with an incidence rate of 22/ 100,000), and in 2003 (1079 cases with an incidence rate of 19.7/ 100,000). In 2007, 778 cases were reported in Jordan with non-meningococcal meningitis, 140 of these cases were from Amman and 490 were from Irbid alone and the rest are from the other parts in Jordan. If we consider as is known that 30% of these infections (non-meningococcal meningitis) are due to S. pneumonia. This means that 233 cases with S. pneumonia meningitis reported annually with 147 from Irbid and 42 cases from Amman which makes 189 cases (81% of all pneumococcal meningitis of Jordan occurring in Irbid and Amman).

Many factors have been identified to promote the clonal spread of multiresistant strains; such as places with high density of children as in DCC and orphanages. S. pneumonia, that are resistant to many antimicrobial agents. Extensive and often excessive use of antibiotics can promote the replacement of strains susceptible to antimicrobial agents by resistant ones (Garcia-Rodriguez and Fresnadillo Martinez 2002), (Pradier, Dunais et al. 1997). Despite adequate antibiotic treatment, morbidity and mortality due to pneumococcal disease remain high (Butler, Shapiro et al. 1999). Moreover, the increase of multidrug resistance among pneumococcal isolates hampers adequate treatment (Crook and Spratt 1998), (Klugman 1996), (Tomasz 1997). These strains are subsequently disseminated in the community by other contacts of colonized children, e.g., their siblings and parents. It is possible to limit the spread of some serotypes of S. pneumoniae by vaccination, but studies of the impact of immunization on colonization have yielded discrepant results (Dagan, Givon-Lavi et al. 2002), (Dagan, Melamed et al. 1996), (Dagan, Muallem et al. 1997), (Mbelle, Huebner et al. 1999). New pneumococcal conjugate vaccines have been shown to be effective against invasive diseases in young children (Black, Shinefield et al. 2000). Furthermore, a protective effect against respiratory tract infections such as (recurrent) otitis media has been observed (Black, Shinefield et al. 2000), (Eskola, Kilpi et al. 2001). Thus far, the 7-valent pneumococcal conjugate vaccine Prevenar (Wyeth) has been approved by the U.S. Food and Drug Administration and the European Committee on Proprietary Medicinal Products and is recommended by the U.S. Advisory Committee on Immunization Practices for the prevention of invasive diseases in children under 2 years of age. Recommendations are also made for older children at increased risk for invasive disease, such as those with human immunodeficiency virus infection and asplenia and those with increased risk for pneumococcal mucosal disease, such as children with recurrent acute otitis media. The effect of the 7-valent pneumococcal conjugate vaccine followed by a 23-valent polysaccharide vaccine in children aged 1 to 7 years with a history of recurrent acute otitis media was studied (Veenhoven, Bogaert et al. 2003). Clinically, no protective effect of the pneumococcal vaccines on recurrence of acute otitis media was found. At the nasopharyngeal level, however, a significant reduction of colonization with vaccine-type pneumococci was found after vaccination, whereas a simultaneous increase in colonization with non vaccine serotypes was observed (Veenhoven, Bogaert et al. 2003), (van der Linden, Al-Lahham et al. 2007). The spread of non-vaccine 19A penicillin resistant pneumococcal strains in the USA is a very serious development indeed, the children had to be treated with levofloxacin and one became partially deaf. With widespread of Prevenar use in Jordan this clone might appear (Pichichero and Casey 2007; Pichichero and Casey 2007). Recently, a Ph D study in Jordan showed that the resistance of penicillin G to S. pneumoniae isolated from healthy children in the kindergarten has reached to 92%. The efficacy of the 7v PCV to define the disease burden in the developing countries has been studied .

SIGNIFICANCE OF WORK

This research project has many dimensions including the following:

* The research project would give an idea about the effect of the vaccine that is given to the children, whether this would affect the incidence of IPD indirectly in the city of Ajlun compared to others.
* As a result of the first point, a governmental National program of vaccination of children will take place for the Jordanian children at specific age
* In addition, the resistance pattern of the isolates against 14 different antibiotics will be developed. High resistance rates will indicate that treatment with such an antibiotic is not efficient and we must use an alternative for the treatment. A precise result of the antibiotic resistance pattern could save money by prescribing antibiotics that are safe and effective, and would educate the Jordanian population about a better use of antimicrobials.
* Furthermore, Serotyping of S. pneumoniae isolates of all pneumococcal strains isolated in this study would give an idea about the coverage of the vaccine available and would answer the families question shall we vaccinate our children or not!! Why should we pay 85 JDs privately to vaccine since the coverage is less than 50% as an example. Here comes the question whether we should use the 13 va,lent vaccine of the same type, which is still under development. Carriage of S. pneumoniae in Jordan pediatrics below 5 was developed in the primary results of the carriage in Jordan and was 57%. if the carriage distribution in the Jordanian population has to do with specific serotypes, which are included in the 7-vPCV, then vaccination would be the best idea to prevent occurrence of the infection then decrease morbidity and later the mortality rate due to the infections of this pathogen. The northern of Jordan constitutes of more than 50% of all non-meningococcal infections.
* An appropriate vaccination program of specific areas and/or specific age groups in Jordan might decrease the distribution of this disease and in turn saving money.
* The results will obtain an insight into the effect of the pneumococcal conjugate vaccine on the genetic pneumococcal population structure.
* The research findings will later on improve the quality of different private and governmental laboratories in Jordan through personal contact and advising. By applying bioinformatics and the phylogeny from the data of resistance, serotyping and Multilocus Sequence Typing (MLST), global clonal relationship of the strains can be obtained from the data.

Study Design: A 15 month surveillance study of Nasopharyngeal Carriage and Antibiotic Resistance of S. pneumoniae in Healthy Jordanian Infants will be launched in Jordan (Ajlun) in the time period between May 2009 to August 2010. Children will be given the 7vPCV as during the 3rd, 5th and 10th months of age (two plus one scheme). Nasopharyngeal swabs will be collected from the DCCs of Ajlun. Questionnaires and special forms will be taken with each isolate and will be sent to the reference lab at the German-Jordanian University for isolation of pneumococci, identification, serotyping, and resistance and for molecular analysis, statistical analysis and coverage. Agreement from the Ministry of Health (MOH), to take all ethical points regarding sample collection into consideration will be guaranteed. The samples will be cultivated at a microbiology lab of the German-Jordanian University. Molecular methods will be investigated in Germany at the National Reference Center for Streptococci. Phases of project implementation will be collection of the samples, and identification.

Culture and identification: Samples will be inoculated on Columbia agar plates with 5% sheep blood. The plates will be incubated at 35°C with 5% CO2 overnight. Identification will be performed by conventional microbiological methods like colony morphology, susceptibility to optochin (bioMérieux), and bile solubility.

Susceptibility testing:

Minimal inhibitory concentration (MIC) testing will be performed using the broth micro broth dilution method recommended by the Clinical Laboratory Standards Institute (CLSI) (CLSI 2008). Antibiotics to be used are Penicillin G, Amoxicillin, Cefotaxime, Cefuroxim, Cefpodoxim, Clarithromycin, Clindamycin, Tetracycline, Levofloxacin, Telithromycin, Trimethoprim/Sulfamethoxazole, Chloramphenicole, Vancomycin and might include other possible new antibiotics as upon request as Tigecycline. S. pneumoniae ATCC 49619 will be included as a control strain.

Analysis of resistance determinants (Geno- and phenotyping): PCR of macrolide resistance determinants will be performed as described previously (Reinert, Lütticken et al. 2003; Reinert 2004; Reinert, Jacobs et al. 2005). For the classical detection of erm(B) and mef(A).

Serotyping:

Pneumococcal strains will be serotyped by Neufeld's Quellung reaction using type and factor sera provided by the Statens Serum Institut, Copenhagen, Denmark.

Subject Population to be Included:

All November 2008 newborns of the Ajlun city (ca 3676/year) - equals 250-300 child/month included in the vaccination program in the time period 1.04.2009 to 28.04.2009 will have Nasopharyngeal swab before the first dose of PCV-7 and a second swab before the third dose at 12th month of age, and a third swab 3 months after the third dose. Swabs will be sent to a reference lab at the German-Jordanian University for identification, serotyping, and resistance testing.

Number of Subjects per Study Group (if applicable): 250-300 infants. Birth cohort in Ajlun is 3676/year representing 250-300 child/month. The study will be conducted on newborns of Jan 2009 coming for the vaccination at their third month of age.

Primary and Secondary Efficacy Endpoints: The frequency of NP carriage, serotype distribution and antimicrobial resistance patterns of the strains in infants less than 2 years old who are not attending daily care centers, who live in rural areas. As there is no truly efficacy in this project, determination and assessment of the reduction in vaccine type pneumococcal carriage as a result of vaccination, so that in this project we will model the impact of a routine program with the 7v PCV based on the serotype coverage in the country. known documented effectiveness in other countries using the same schedule, since it is well known that the 7v PCV can prevent. Rate of resistant strains.

Statistical Considerations: Statistical analysis will be done after completion of the project, epidemiological statistics including: Calculate the percentage of Nasopharyngeal Carriage with vaccine type and non vaccine type at each time of isolation from each newborn, resistance to antibiotics (percentage of resistance, MIC50, MIC90 and range): demographic analysis for age, sex, and others like presence of a child within the house who attends school, socio-economical level, antibiotic use before the last 30 days, sleeping room- alone or with siblings and presence of a smoker in the house.

Institutional Review Board (IRB)/Independent Ethics Committee (IEC) Approval: Include information about the IRB/IEC, confirming that its composition and mechanism for provision of approval are consistent with International Conference on Harmonization, Food and Drug Administration (FDA) Code of Federal Regulations (CFR), and/or local and regional requirements and that all necessary IRB/IEC approval and Competent Authority approvals will be obtained in connection with the proposed research.

Informed Consent/Privacy Authorization: Include information on the manner in which informed consent is obtained and adherence to applicable regulations including applicable privacy regulations.

All enrolled infants in the daily care centers, the parents or the mother or father would be respectfully asked to sign a document of agreement for the vaccination with the 7v PCV, and to take NP swabs from the infants enrolled, and to take data for protocoling and those parents will be educated on the benefits of the vaccination before vaccination.

Phase 1: Started in June 2009 to August 2009, with collection of 377 NP-samples from 2 months age infants after the first injection with 7v PCV in Ajlun. As a result 133 strains of Streptococcus pneumoniae were isolated.

ELIGIBILITY:
Inclusion Criteria:

* All infants who were enrolled in the time period May 18th, 2009 to August 10th, 2010, would have the 7v PCV
* Those infants who have no exclusion criteria

Exclusion Criteria:

* Isolates from the same patient as duplicates will not be considered

Ages: 2 Months to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 377 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-08 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Decrease colonization with S. pneumoniae. | 1.5 years maximum

SECONDARY OUTCOMES:
Decrease infections related to S. pneumoniae by infants and indirectly elderly of same families and decrease use of Antibiotics and therefore the resistance | 1.5 years to finish the whole trial

CONTACTS AND LOCATIONS:
Overall Officials: Adnan AL-lahham, PhD, Principal Investigator — German Jordanian University/ School of Applied Medical Sciences/ P.O.Box 35247 Amman/ 11180 Amman, Jordan
Locations (1):
- German Jordanian University, Amman, Amman Governorate, Jordan